CLINICAL TRIAL: NCT06193239
Title: Diagnostic Accuracy Study for OWL-EVO1 As a Lung Cancer EVOC® Probe
Brief Title: Diagnostic Accuracy Study for OWL-EVO1 As a Lung Cancer EVOC® Probe (Evolution Phase 2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Owlstone Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OML-EV2-1.0
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Diagnostic Test; Diagnostic Breath test
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants with and without suspicion of having lung cancer will all receive the same IMP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OWL-EVO1 (Experimental): After confirming full eligibility, individuals will all be administered the OWL-EVO1 probe intravenously.
  This includes:
  * Patients diagnosed with histopathologically confirmed lung cancer.
  * Individuals with a CT-proven absence of lung cancer, including those with relevant comorbidities and risk factors such as smoking, COPD, asthma, extrapulmonary malignant tumours, active lung infection/inflammation and other chronic respiratory diseases.
  Interventions: Diagnostic Test: OWL-EVO1

INTERVENTIONS:
Diagnostic Test: OWL-EVO1 — EVOC probe
  Other Names: OWL-EVO1 Breath Biopsy Test; D5-ethyl-βD-glucuronide

SUMMARY:
The Phase 2a Evolution study aims to assess the diagnostic accuracy of the OWL-EV1 Probe Breath Biopsy Test to differentiate between individuals with lung cancer and relevant contrast groups.

The contrast groups will be representative of the clinical populations in which the test is intended to be used.

Thus, Evolution Phase 2a will be designed as a cross-sectional, case-control trial that will be conducted at various sites, both in the UK and EU.

DETAILED DESCRIPTION:
In Evolution Phase 1, Owlstone Medical demonstrated the safety and tolerability of their Exogenous Volatile Organic Compound (EVOC) Probe. This phase also demonstrated proof of mechanism for the cleavage of the EVOC Probe, D5-ethyl-βD-glucuronide (OWL-EVO1), into D5-ethanol which can be detected on breath. This makes OWL-EVO-1 a promising EVOC Probe for the detection of lung cancer.

The Evolution Phase 2a study will evaluate the diagnostic accuracy of an OWL-EVO1 based breath test for the differentiation of those with histopathologically confirmed lung cancer and relevant contrast groups with a CT-proven absence of lung cancer. These contrast groups will include those with relevant comorbidities, to truly evaluate accuracy and the robustness of test performance.

As a secondary objective, the study aims to define a test protocol that minimises healthcare worker effort, whilst maximising tolerability and diagnosed accuracy for the intended use setting.

This phase intends to recruit up to 150 cases and 200 controls. Both cohorts will be administered the probe intravenously. Multiple breath samples will be collected for up to 180 minutes post-probe infusion, with the cumulative sampling time not exceeding 60 minutes.

The study results will provide valuable insights into the expected test performance as well as optimisation of the test in a clinical pathway.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-85 years.
* Ability to provide informed consent.
* BMI 16 - <40.
* Receiving a CT including the thoracic region, within the last 6 months.

Exclusion Criteria:

1. (Anticipated) inability to complete the breath sampling procedure (e.g., inability to maintain adequate ventilation unaided or claustrophobia).
2. Potential subjects who in the opinion of the investigator lack mental capacity.
3. Received an investigational medical product in the context of a Clinical Trial (CTIMP) during the 28 days prior to administration of the (first) probe, or within 5 times the half-life of the investigational medicinal product previously received, whichever is longer.*
4. Individuals under diagnostic investigation for a potential malignancy other than lung cancer that has not yet reached a conclusive diagnosis**.
5. Individuals with an inconclusive lung abnormality (indeterminate pulmonary nodule) on CT-scan requiring CT-based monitoring rather than biopsy and/or treatment.
6. Documented history of pulmonary surgery or endobronchial interventional procedures other than biopsy, lavage, or bronchial brushings. These include surgical resection, Video Assisted Thoracic Surgery (VATS), bronchial thermoplasty and coiling, airway stenting or other interventional bronchoscopic procedures.
7. Pregnant or breastfeeding women and women of child-bearing potential not using adequate contraceptive methods (Subjects must agree to use contraception for 2 months post last dose).
8. Individuals under investigation for suspicion of lung cancer who are unlikely to receive a definitive tissue diagnosis of lung cancer prior to treatment (e.g. stereotactic ablative radiotherapy without tissue confirmation).

   * Note:

In the case that the participant has taken part in a study with an investigational medicinal product please contact the Owlstone medical monitor for advice.

**Note: Individuals with a confirmed cancer diagnosis ARE eligible (such as a diagnosis of prostate cancer now undergoing hormone therapy). Individual with a previous history of cancer other than lung cancer, including those under active surveillance, ARE eligible. Individuals scheduled to attend a cancer screening program; prostate, breast, lung, colon, ARE eligible.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 12 months
  The primary endpoint is to assess the diagnostic accuracy of the OWL-EVO1 Breath Biopsy test to differentiate between individuals with lung cancer and contrast groups. This will be reported using a Receiver Operator Characteristic Curve, NPV, PPV, Sensitivity, Specificity & Likelihood Ratio's. Metrics will be reported for overall test performance as well as pre-defined subgroup analyses.

SECONDARY OUTCOMES:
Optimised test | 12 months
  To define a test protocol for breath sampling and the OWL-EVO-1 infusion that achieves the optimal balance between minimising healthcare worker effort, maximising tolerability, and optimising diagnostic accuracy for the intended use setting. This will be in terms of method, timing, posture and duration.
Safety and tolerability | 12 months
  To gain a refined understanding of the safety and tolerability of OWL-EVO1. This will be based on reported Adverse Events associated with probe administration.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rintoul, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust
Locations (9):
- Thomayer Hospital, Prague, Prague, Czechia
- Hungary (2):
  - National Koranyi Institute for Pulmonology, Budapest, Budapest
  - Department of Pulmonology, University of Debrecen, Debrecen, Debrecen
- United Kingdom (6):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Wythenshawe Hospital, Manchester, Greater Manchester
  - Glenfield Hospital, Leicester, Leicestershire
  - Barts Health NHS Trust, London, London
  - Imperial Centre for Translational and Experimental Medicine, Imperial College, London, London
  - Quadram Institute, Norwich, Norfolk

IPD SHARING:
Plan to Share IPD: No